CLINICAL TRIAL: NCT01050985
Title: A Phase I Study of the mTOR Inhibitor Temsirolimus Plus Capecitabine in Patients With Advanced Malignancies
Brief Title: A Study of Temsirolimus Plus Capecitabine in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-479
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Advanced Solid Tumors
Keywords: advanced cancer; temsirolimus; capecitabine
MeSH Terms: interventions — temsirolimus; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- temsirolimus and capecitabine (Experimental): Treatment with the combination of temsirolimus and capecitabine
  Interventions: Drug: Temsirolimus and capecitabine

INTERVENTIONS:
Drug: Temsirolimus and capecitabine — temsirolimus in escalating doses starting at 15-mg IV on days 1 and 8 of a 14 day cycle capecitabine in escalating doses starting at 1000 mg/m2 by mouth twice a day on days 1-7 of a 14-day cycle
  Other Names: Temsirolimus; Torisel; CC-779; NSC 022088; Capecitabine; Xeloda

SUMMARY:
This study is for people with advanced cancer for which no curative treatment exists.

The purpose of this study is to test the safety and effectiveness of the combination of the drugs Temsirolimus and Capecitabine and see what effects it has on cancer.

Temsirolimus is a drug that is given by vein that targets a protein important for the growth of cancer cells known as mTOR. By inhibiting this protein, Temsirolimus can inhibit cancer cell growth and even lead to their death.

Capecitabine is a more traditional chemotherapy. It is an oral pill that gets converted in the body to the very common chemotherapy known as 5-fluorouracil.

This research is being done because it is not known if the combination of Temsirolimus and Capecitabine will work better than Capecitabine or Temsirolimus alone.

DETAILED DESCRIPTION:
This is a Phase I study designed to assess the safety and clinical activity of temsirolimus in combination with capecitabine in patients with advanced malignancies. Because the toxicities of capecitabine are well established, and based on a previous clinical trial of temsirolimus and continuous infusion 5-fluorouracil, an alternating dose escalation plan will be employed.

The first stage of the study will be performed to identify the maximally tolerated dose of the combination, when capecitabine is given on a every 2 week schedule. The starting dose of temsirolimus will be 15-mg IV on day 1 and 8 plus capecitabine 1000 mg/m2 by mouth twice a day on days 1-7 of a 14 day schedule. Patients will be enrolled in a standard 3+3 dose escalating fashion to a maximum dose of temsirolimus of 25-mg and a maximum dose of capecitabine of 1750 mg/m2 twice a day.

If the maximally tolerated dose is determined for the every 2 week schedule, then in the second stage of the study a similar dose escalation plan will be employed for an every 3 week schedule.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma with measurable or evaluable disease
* Disease for which capecitabine is approved or compendia listed
* Advanced unresectable, and/or metastatic disease for which there is no known curative therapy
* Performance status 0-2
* Adequate hepatic, bone marrow, and renal function

Exclusion Criteria:

* Brain metastases not under control for at least 3 months
* Active severe infection or known chronic infection with HIV, hepatitis B virus, or hepatitis C virus
* Cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia, or myocardial infarction, stroke, or congestive heart failure within the last 6 months
* Life-threatening visceral disease or other severe concurrent disease
* Women who are pregnant or breastfeeding
* Anticipated patient survival under 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Identification of the recommended Phase II dose of temsirolimus to be used in combination with capecitabine in patients with advanced malignancies | 1 year

SECONDARY OUTCOMES:
Evaluation of toxicity of the combination of temsirolimus plus capecitabine in patients with advanced malignancies as determined by adverse events observed and lab values | 1 year
To determine the response by radiology scans to temsirolimus and 5-FU-based therapies in patients with advanced malignancies | 9 weeks
Comparison of the response rate in patients whose tumors demonstrate activation of the mTOR pathway versus those that do not | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Pishvaian, Md, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States